CLINICAL TRIAL: NCT06107530
Title: Living a Pregnancy After a Peri-natal Grief: How Well Does Pregnancy Follow-up Meet Women's Needs and Expectations?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GARDEN
Record Dates: First submitted 2023-10-05; First posted 2023-10-30 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Pregnancy Related
Keywords: peri-natal loss; pregnancy follow up

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Semi structured interview (Experimental)
  Interventions: Other: semi structured interview

INTERVENTIONS:
Other: semi structured interview — Women fulfilling the inclusion / exclusion criteria will be asked to participate to a semi structured interview with a psychiatrist or a psychologist

SUMMARY:
Every year in France, around 7,000 children are born without life, following a medical termination of pregnancy (IMG), fetal death in utero (FDIU) or premature delivery ("late miscarriage"). For families affected by perinatal bereavement, the pregnancy that follows this silent birth is a moment apart, between anguish and guilt, joy and apprehension. The aim of this research project is to improve the understanding of what women go through during the pregnancy that follows, with a view to proposing a practical tool for the professionals who take care of them, in order to improve and personalize their follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Women who have given birth to a stillborn child (singleton or twin pregnancies):

  * delivery following fetal death in utero or medical termination of pregnancy at 15 weeks gestational age and later
  * extreme preterm birth ("late miscarriage") from 15 weeks gestational age Patient who subsequently carried a pregnancy to term and gave birth to a live, viable child between 2020 and 2023.
* French-speaking patient
* Patient who does not object to her participation in this research study

Exclusion Criteria:

* Women who have experienced a natural termination of pregnancy ("early miscarriage") before 15 weeks of amenorrhea.
* Women who have given birth by suction in the operating theatre.
* Women who are pregnant with twins in the pregnancy following bereavement. Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Identify women's specific needs and expectations for the follow-up of this particular pregnancy | 4months

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation hôpital Saint Joseph, Paris, France

IPD SHARING:
Plan to Share IPD: No